CLINICAL TRIAL: NCT05627323
Title: A Phase 1b Study to Evaluate CHM-1101, a CAR T-Cell Therapy With a Chlorotoxin Tumor-Targeting Domain for Patients With Matrix Metallopeptidase 2 Positive (MMP2+) Recurrent or Progressive Glioblastoma Multiforme
Brief Title: CAR T Cells in Patients With MMP2+ Recurrent or Progressive Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chimeric Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-1101-001
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: Progressive or recurrent glioblastoma; MMP2+
MeSH Terms: conditions — Glioblastoma | interventions — Chlorotoxin

STUDY DESIGN:
Intervention Model Description: Two dose levels investigated, with both dose levels proceeding in parallel. Expansion or de-escalation decision rules are based on a traditional 3+3 clinical study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (CAR T cell therapy) 1 (Experimental): Arm 1 participants will undergo resection of their tumor. Participants receive half the CHM-1101 dose via Rickham catheters into the tumor cavity and half into the lateral ventricle.
  Cycle 1 (28 days) CHM 1101 total dose will be divided across 3 once-weekly administrations.
  After Cycle 1, additional cycles may be initiated in the absence of disease progression or unacceptable toxicity provided that the principal investigator and participant agree to continue and if adequate autologous CAR-T doses remain.
  Interventions: Biological: CHM-1101 CAR-T cells
- Treatment (CAR T cell therapy) 2 (Experimental): Arm 2 participants will undergo resection of their tumor. Participants receive half the CHM-1101 dose via Rickham catheters into the tumor cavity and half into the lateral ventricle.
  Cycle 1 (28 days) CHM 1101 total dose will be divided across 3 once-weekly administrations.
  After Cycle 1, additional cycles may be initiated in the absence of disease progression or unacceptable toxicity provided that the principal investigator and participant agree to continue and if adequate autologous CAR-T doses remain.
  Interventions: Biological: CHM-1101 CAR-T cells

INTERVENTIONS:
Biological: CHM-1101 CAR-T cells — Administered via ICT/ICV dual delivery
  Other Names: Chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes (via ICT/ICV dual delivery); Chlorotoxin-CD28-CD3z-CD19t-expressing CAR T-cells

SUMMARY:
This is a phase 1b study to evaluate the safety of chimeric antigen receptor (CAR) T cells with a chlorotoxin tumor-targeting domain (ie, CHM-1101, the study treatment) to determine the best dose of CHM-1101, and to assess the effectiveness of CHM-1101 in treating MMP2+ glioblastoma that has come back (recurrent) or that is growing, spreading, or getting worse (progressive).

DETAILED DESCRIPTION:
This is a phase 1b, multicenter, feasibility/safety study of the dual delivery (administered through both intracavitary/intratumoral [ICT] and intraventricular [ICV] catheters) of CHM-1101, an autologous chlorotoxin-chimeric antigen receptor (CLTX-CAR) cell product, in participants with recurrent or progressive GBM. The investigational product is identified as CHM-1101 (CLTX(EQ)28ζ/CD19t+ CAR T cells).

PRIMARY OBJECTIVE

• To determine the recommended phase 2 dose (RP2D) for dual ICT and ICV delivery of CHM-1101 in participants with MMP2+ recurrent or progressive GBM.

SECONDARY OBJECTIVES

* To assess the feasibility and safety of dual delivery of CHM-1101.
* To describe the persistence, expansion, immunogenicity, and phenotype of CHM-1101 and endogenous cells tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF).
* In participants who receive at least 2 of the 3 planned doses of CHM-1101 in Cycle 1:

  * Estimate the progression-free survival (PFS) rates
  * Estimate the overall survival (OS) rates
* To evaluate the disease response rate.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the subject and/or legally authorized representative.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.
* Age 18 years and older.
* ECOG status of 0 or 1.
* Life expectancy ≥12 weeks.
* Subject has a prior histologically confirmed diagnosis of a grade 4 glioblastoma multiforme (GBM) or a prior histologically confirmed diagnosis of a grade 2 or 3 malignant glioma and now has radiographic progression consistent with a grade 4 GBM (IDH wild type), grade 4 diffuse astrocytoma (IDH mutant), or has a unifocal relapse of GBM.
* Relapsed disease: radiographic evidence of recurrence/progression of measurable disease after standard therapy and ≥ 12 weeks after completion of front-line radiation therapy.
* Confirmed MMP2+ tumor expression by IHC (≥20% moderate/high MMP2 score [2+ or 3+]).
* Adequate venous access to perform leukapheresis.
* No known contraindications to leukapheresis or steroids.
* In-range baseline laboratory values for WBC (>2000/dL [or ANC ≥1000/mm^3]), platelets (≥75000/mm^3), total bilirubin (≤1.5xULN), AST (≤2.5xULN), ALT (≤2.5xULN), serum creatinine (≤1.5xmg/dL), and oxygen saturation (≥95% on room air)
* Seronegative for human immunodeficiency virus (HIV) by antigen/antibody (Ag/Ab) testing.
* Seronegative for hepatitis B and/or hepatitis C virus.
* Women of childbearing potential must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
* Agreement by women AND men of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of CHM-1101. (Childbearing potential is defined as not being surgically sterilized (women and men) or, for women, having not been free from menses for > 1 year.)

Exclusion Criteria:

* Within 3 months of having received prior bevacizumab therapy at the time of enrollment.
* Not yet recovered from toxicities of prior therapy.
* Uncontrolled seizure activity and/or clinically evident progressive encephalopathy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Clinically significant uncontrolled illness.
* Active infection requiring antibiotics.
* Known history of HIV or hepatitis B or hepatitis C infection.
* Other active malignancy.
* Women only-pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective subjects who, in the opinion of the Investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2041-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Cytokine Release Syndrome (CRS) | up tp 15 years
  Assessed per American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading guideline, evaluating levels and phenotype detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) (absolute number per µL by flowcytometry).
All other adverse events and toxicities | up to 15 years
  Assessed per NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Chimeric antigen receptor (CAR) T cell | up to 15 years
  Assess levels and phenotype detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) (absolute number per µL by flowcytometry).
Endogenous T cell | up to15 years
  Assess level and phenotype detected in TCF, PB, and CSF (absolute number per µL by flowcytometry).
Human anti-CAR antibody (HACA) | up to 15 years
  Serum samples will be evaluated for HACA against the CLTX(EQ)28ζ therapeutic agent.
Progression free survival (PFS) time | 12 months
  Measured from the date of first infusion of CAR-T cells until the first date when progressive disease (PD) is objectively documented or death from any cause, whichever is earlier.
Overall survival (OS) | up to 15 years
  Measured from the date of first infusion of CAR-T cells until death.
Disease response | 12 months
  Assessed by modified Response Assessment in Neuro-Oncology Criteria (RANO) criteria.
Clinical benefit rate | 12 months
  The proportion of participants who experience a complete response, a partial response, or stable disease that is 3 months or greater in duration.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - St. David's South Austin Medical Center - Sarah Cannon - Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No